CLINICAL TRIAL: NCT03417583
Title: Assessing Efficacy of Neuropsychiatric Assessment and Treatment Protocols in Huntington's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Principal Investigator, David Isaacs, Movement Disorder Fellow, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 172030
Record Dates: First submitted 2018-01-23; First posted 2018-01-31 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Standard Care Group (No Intervention): These patients will continue to be seen by their regular neurology provider for Huntington's disease. They will not be treated explicitly according to the protocol, though they may be prescribed some of the same medications.
- Protocol Intervention Group (Experimental): These participants will transfer their clinical care to the study provider for the duration of the study, and their symptom treatment will be guided by the study protocol.
  Interventions: Other: Protocol Intervention Group

INTERVENTIONS:
Other: Protocol Intervention Group — For neuropsychiatric symptoms identified by the clinician, the treatment protocol, based on clinical standard of care, will be implemented. This protocol includes directions for multidisciplinary treatment of 7 neuropsychiatric symptoms: depression, apathy, anxiety, agitation/irritability, obsessive compulsive behaviors, delusions/hallucinations, and sleep dysfunction. These treatment recommendations differ according to symptom but include provision of additional information to patients and caregivers, psychotherapy/counseling, and pharmacotherapeutic treatment options including recommended agents and follow-up schedule.
  Arms: Protocol Intervention Group

SUMMARY:
Phase A: Recruit 50 patients with HD, and their caregivers, to complete a neuropsychiatric and quality of life battery of scales at baseline. Have these 50 patients complete a formal psychiatric assessment with a psychiatrist within 2 weeks of this clinical battery, and the results of these 2 types of assessments will be compared to establish the level of agreement between clinical rating scales and formal psychiatric assessment.

Phase B: Continue to follow Phase A cohort longitudinally and administer neuropsychiatric and quality of life battery at 6 months, 12 months, and 18 months form baseline. Recruit an additional 50 patients, administer the same neuropsychiatric and quality of life battery at baseline, implement medication and counseling intervention according to a standard of care protocol, and follow up with the same neuropsychiatric and quality of life battery at 6, 12, and 18 months.

DETAILED DESCRIPTION:
As presented to Phase A (control) patient participant:

"If you are in this study, you will be asked to answer a series of online surveys assessing your psychiatric symptoms and quality of life in the presence of a caregiver. These surveys will be emailed to your consented caregiver in the week before your in-person visit. You will then come to clinic for an in-person assessment of psychiatric and motor symptoms of HD. You will also undergo an in-person psychiatric evaluation with a psychiatrist at Vanderbilt who works with HD patients. This psychiatric evaluation will take approximately 60 minutes and will occur up to 2 weeks before or after your first regular study visit. This involves a clinical interview during which a psychiatrist, who is an expert in psychiatric symptoms of HD, will ask about your experience with many different symptoms that can be experienced in HD. These two in-person evaluations will occur within 2 weeks of each other. You will continue to see your neurology provider for routine follow-up, and you will return for in-person follow-up assessments at 6 months, 12 months, and 18 months, repeating the online surveys prior to each visit.

Health-Related Quality of Life and Psychiatric Symptom Surveys (This will take approximately 60-90 minutes):

You will be asked to answer on-line survey questions about your psychiatric symptoms and quality of life in the presence of a caregiver.

* The Neuro-QoL scales include 4 subscales created specifically to measure quality of life in patients with neurological disease. These scales include 33 total questions which ask you to report your anxiety, depression, sense of well-being, and satisfaction with social roles within the previous week.
* The PROMIS Anger scale includes 8 questions that ask you to rate your symptoms of anger in the previous week.
* The PROMIS Sleep-Related Impairment short form includes 8 questions that ask about your sleep quality and how you feel during the day after sleeping.
* The Patient Health Questionnaire- 9 (PHQ-9) includes 9 questions about symptoms of depression that you may be experiencing and how these affect you on a daily basis.
* The HD Anosognosia Rating Scale includes 8 questions that ask you to assess how you perform daily tasks compared to other people of your same age and education level.
* Sleep Questionnaire includes 5 questions about your night and daytime sleep habits.
* We will also gather background information such as: date of birth, where you live, if you have insurance, and your income. You will also be asked about health and medical history such as: when you were diagnosed with HD and what medications you are taking.

Psychiatric and Motor Symptom Assessment (This will take approximately 60 minutes):

* The Hamilton Anxiety Rating Scale (HAM-A) asks you to rate the severity of 14 anxiety symptoms.
* The Problem Behaviors Assessment short form (PBA-s) asks you and your caregiver about the frequency and severity of 11 different psychiatric symptoms that can be experienced in HD.
* The Columbia Suicide Severity Rating Scale includes up to 6 items yes or no questions to assess presence and severity of suicidal thoughts.
* The Montreal Cognitive Assessment (MOCA) is short test to measure your memory and thinking skills.
* The United Huntington's Disease Rating Scale (UHDRS) tool is used by HD clinicians to measure the presence and severity of your motor symptoms like chorea and walking difficulty.
* The UHDRS Total Functional Capacity (TFC) scale is used by HD clinicians to rate your ability to carry out daily tasks such as household chores or managing finances."

As presented to Phase B (protocol) patient participant:

"If you are in this study, you will be asked to answer a series of online surveys assessing your psychiatric symptoms and quality of life in the presence of a caregiver. These surveys will be emailed to your consented caregiver in the week before your in-person visit. You will then come to clinic for an in-person assessment of psychiatric and motor symptoms of HD. In addition, your psychiatric symptoms will be treated according to a systematic protocol developed by HD experts that guides treatment decisions based on our current clinical standard of care. You will return for in-person follow-up assessment at 6 months, 12 months, and 18 months, repeating the online surveys prior to each visit.

Health-Related Quality of Life and Psychiatric Symptom Surveys (This will take approximately 60-90 minutes):

You will be asked to answer on-line survey questions about your psychiatric symptoms and quality of life in the presence of a caregiver.

* The Neuro-QoL scales include 4 subscales created specifically to measure quality of life in patients with neurological disease. These scales include 33 total questions which ask you to report your anxiety, depression, sense of well-being, and satisfaction with social roles within the previous week.
* The PROMIS Anger scale includes 8 questions that ask you to rate your symptoms of anger in the previous week.
* The PROMIS Sleep-Related Impairment short form includes 8 questions that ask about your sleep quality and how you feel during the day after sleeping.
* The Patient Health Questionnaire- 9 (PHQ-9) includes 9 questions about symptoms of depression that you may be experiencing and how these affect you on a daily basis.
* The HD Anosognosia Rating Scale includes 8 questions that ask you to assess how you perform daily tasks compared to other people of your same age and education level.
* Sleep Questionnaire includes 5 questions about your night and daytime sleep habits.
* We will also gather background information such as: date of birth, where you live, if you have insurance, and your income. You will also be asked about health and medical history such as: when you were diagnosed with HD and what medications you are taking.

Psychiatric and Motor Symptom Assessment (This will take approximately 60 minutes):

* The Hamilton Anxiety Rating Scale (HAM-A) asks you to rate the severity of 14 anxiety symptoms.
* The Problem Behaviors Assessment short form (PBA-s) asks you and your caregiver about the frequency and severity of 11 different psychiatric symptoms that can be experienced in HD.
* The Columbia Suicide Severity Rating Scale includes up to 6 items yes or no questions to assess presence and severity of suicidal thoughts.
* The Montreal Cognitive Assessment (MOCA) is short test to measure your memory and thinking skills.
* The United Huntington's Disease Rating Scale (UHDRS) tool is used by HD clinicians to measure the presence and severity of your motor symptoms like chorea and walking difficulty.
* The UHDRS Total Functional Capacity (TFC) scale is used by HD clinicians to rate your ability to carry out daily tasks such as household chores or managing finances."

As presented to caregiver participant:

"If you are involved in this study, you will be asked to assist the HD patient in completing a series of online surveys assessing his or her psychiatric symptoms and quality of life. You will also be asked to complete an online survey about your experience as a caregiver:

• The Traumatic Brain Injury- Care Quality of Life (TBI-CareQOL) Caregiver Strain short form includes 6 items which ask you to rate your feelings of stress and strain related to being a caregiver.

All surveys will be emailed to you the week prior to an in-person study visit.

You will then accompany the HD patient to clinic for an in-person assessment of psychiatric and motor symptoms of HD. During this visit you will be asked to answer questions about the patient's psychiatric symptoms (see scales below) and offer input on other symptom surveys directed to the patient as you would in a normal clinic visit.

* The Factor analysis of the frontal systems behavior scale (FrSBe) family-version is a 46-item scale that asks you to rate characteristics of frontal lobe dysfunction that you observe in the HD patient currently and prior to disease onset.
* The Problem Behaviors Assessment short form (PBA-s) asks you and the HD patient about the frequency and severity of 11 different psychiatric symptoms that can be experienced in HD. "

ELIGIBILITY:
Inclusion Criteria:

Patient participants:

* Diagnosed with HD, either through genetic testing or neurologist's clinical diagnosis
* Patient has at least 1 neuropsychiatric symptom, as reported by their HD provider
* 21 and older will be included, as symptoms of Juvenile HD (in patients 20 years old or less) can present differently
* Presence of an eligible caregiver who can also participate in the study with them because several of the study measures require caregiver report

Caregivers:

* 18 years or older
* A caregiver will be defined as someone who lives with or has at least weekly contact with the HD patient

Exclusion Criteria:

Patient participants:

* 20 years old or younger
* Greater than moderate impairment on dementia screening
* Lack of a caregiver to provide collateral information and complete caregiver assessments will also be excluded

Caregivers:

* Younger than 18 years old and/or have less than weekly contact with the HD patient
* Clinical impression of incompetency to answer survey questions as determined by the Jessie Sellers, Nurse Practitioner, or the neurologist caring for the HD patient, then he or she will not be eligible to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Change in quality of life- Concern with Death and Dying | Baseline to 18 months
  This is measured using the HDQLIFE Concern with Death and Dying scale, which measures concern with death and dying in Huntington's disease patients. The total score will range from 6 to 30, with higher scores indicating greater concern with death and dying.
Change in quality of life- Meaning and Purpose | Baseline to 18 months
  This is measured using HDQLIFE Meaning and Purpose scale, which measures feelings of meaning and purpose in Huntington's disease patients. The total score will range from 4 to 20, with higher scores indicating greater feelings of meaning and purpose in life.
Change in quality of life- Ability to Participate in Social Roles and Activities | Baseline to 18 months
  This is measured using the NeuroQoL- Ability to Participate in Social Roles and Activities scale, which measures ability of individuals with neurological conditions to participate in social roles and activities. The total score will range from 8 to 40, with higher scores indicating greater ability to participate in social roles and activities.
Change in quality of life- Anxiety | Baseline to 18 months
  This is measured using the NeuroQoL- Anxiety scale, which measures anxiety in individuals with neurological conditions. The total score will range from 8 to 40, with higher scores indicating greater levels of anxiety.
Change in quality of life- Depression | Baseline to 18 months
  This is measured using the NeuroQoL- Depression scale, which measures depression in individuals with neurological conditions. The total score will range from 8 to 40, with higher scores indicating greater levels of depression.
Change in quality of life- Positive Affect and Well-Being | Baseline to 18 months
  This is measured using the NeuroQoL- Positive Affect and Well-Being scale, which measures positive affect and sense of well-being in individuals with neurological conditions. The total score will range from 9 to 45, with higher scores indicating a greater sense of well-being.
Change in quality of life- Satisfaction with Social Roles and Activities | Baseline to 18 months
  This is measured using the NeuroQoL- Satisfaction with Social Roles and Activities scale, which measures satisfaction with social roles and activities in individuals with neurological conditions. The total score will range from 8 to 40, with higher scores indicating greater levels of satisfaction with social roles and activities.
Change in quality of life- Caregiver Strain | Baseline to 18 months
  This is measured using the TBI-CareQoL- Caregiver Strain scale, which measures health related quality of life in caregivers. The total score will range from 6 to 30, with higher scores indicating greater levels of caregiver strain.

CONTACTS AND LOCATIONS:
Overall Officials: David Isaacs, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided